CLINICAL TRIAL: NCT02134613
Title: 99mTc-anti-TNF-alpha Scintigraphy in the Evaluation of Inflammatory Processes Activity
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, Bianca Gutfilen, Associate Professor, Universidade Federal do Rio de Janeiro
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CONEP-711/2008
Record Dates: First submitted 2014-04-28; First posted 2014-05-09 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-05

CONDITIONS: Psoriatic Arthritis; Arthritis
Keywords: 99mTc-anti-TNF; Inflammation; Psoriatic arthritis; Rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Psoriatic; Arthritis; Inflammation; Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- anti-TNF-alpha scintigraphy (Experimental): 99mTc-anti-TNF-alpha Scintigraphy will be compared with MRI results, analysed and discussed by physicians who are in charge of the patients.
  Interventions: Other: 99mTc-anti-TNF-alpha Scintigraphy

INTERVENTIONS:
Other: 99mTc-anti-TNF-alpha Scintigraphy — 99mTc-anti-TNF-alpha Scintigraphy will be analysed and discussed by physicians who are in charge of the patients.

SUMMARY:
Rheumatoid and psoriatic arthritis patients benefit from anti-TNF-α therapy, once it is effective in reducing joint and skin manifestations in 60-70% of patients with inflammatory articular joint and skin diseases. Thus, identifying the presence and amount of TNF-α in the joint or skin in these patients may help in guiding the course of treatment more efficiently. The investigators research group has developed a novel approach to label anti-TNF-α with technetium-99m. Here the investigators compare the results obtained with scintigraphy and MRI in rheumatoid and psoriatic arthritis. The 99mTc-anti-TNF-α scintigraphy might recognize the molecule involved in the inflammatory process and provide crucial information to help physicians taking decisions about the drugs to be used based on biological evidence and which are cost-effective and appropriate for the treatment of choice. It allows direct identification of the monoclonal antibody anti-TNF-α in the articular joints and skin while it also ensures that the drug has reached its therapeutic target. It also allows correlation between the presence of the drug and clinical responses.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid Arthritis (RA) patients must have 1 joint with edema.
* Inflammatory lumbalgia
* ankylosing spondylitis
* Psoriatic arthritis with active disease and skin lesion

Exclusion Criteria:

* Patients that do not return to scintigraphy
* Pregnancy, Lactation, active infection, severe concomitant disease and medication allergy history

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-01; Primary Completion 2017-07 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with 99mTc-anti-TNF-alpha joint and skin uptake | 1 week

SECONDARY OUTCOMES:
Percentage of Participants with decreased 99mTc-anti-TNF-alpha uptake after follow-up | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Bianca Gutfilen, PhD, Principal Investigator — UFRJ
Locations (1):
- Hospital Universitário Clementino Fraga Filho, Rio de Janeiro, Rio de Janeiro, Brazil

REFERENCES:
- [Derived] Alexandre DJA, Carmo CCM, Romeiro LD, Gutfilen-Schlesinger G, Amarante JLM Jr, de Souza SAL, Gutfilen B. 99mTc-antitumor necrosis factor-alpha scintigraphy for the detection of inflammatory activity in rheumatoid arthritis. Nucl Med Commun. 2021 Apr 1;42(4):389-395. doi: 10.1097/MNM.0000000000001333. PMID 33306625